CLINICAL TRIAL: NCT01325298
Title: UVA-Riboflavin Crosslinking Treatment of Corneal Ectasia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mercy Center for Corrective Eye Surgery (Other)
Responsible Party: Robert L. Epstein, MD, Mercy Center for Corrective Eye Surgery
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IND 109752
Record Dates: First submitted 2011-03-28; First posted 2011-03-29 (Estimated); Last update posted 2011-03-29 (Estimated); Status verified 2011-03

CONDITIONS: Keratoconus; Ectasia; Corneal Ectasia
Keywords: Keratoconus; Ectasia; cross linking; collagen cross linking; corneal crosslinking; corneal diseases; eye diseases
MeSH Terms: conditions — Keratoconus; Dilatation, Pathologic; Corneal Diseases; Eye Diseases | interventions — Riboflavin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 20 Minute UV-X Light Treatment Duration (Active Comparator): 20 Minute UV-X Light Treatment Duration
  Note: "UV-X" is the trademark of Peschke GmbH
  Interventions: Device: UV-X Light; Drug: Riboflavin
- 30 Minute UV-X Light Treatment Duration (Active Comparator): 30 Minute UV-X Light Treatment Duration
  Interventions: Device: UV-X Light; Drug: Riboflavin

INTERVENTIONS:
Device: UV-X Light — UV-X 365 nm wavelength light source is applied to the cornea with continued application of riboflavin 0.1%
  Arms: 20 Minute UV-X Light Treatment Duration
Drug: Riboflavin — Riboflavin 0.1% is applied to the cornea every 2 minutes for 14 minutes prior to and also during UV-X Light treatment.
  Arms: 20 Minute UV-X Light Treatment Duration
Device: UV-X Light — UV-X 365 nm wavelength light source is applied to the cornea with continued application of riboflavin 0.1%
  Arms: 30 Minute UV-X Light Treatment Duration
Drug: Riboflavin — Riboflavin 0.1% is applied to the cornea every 2 minutes for 14 minutes prior to and also during UV-X Light treatment.
  Arms: 30 Minute UV-X Light Treatment Duration

SUMMARY:
The primary objective of this study is to evaluate two different ultraviolet (UV) dosing regimens for corneal collagen cross linking to slow the progressive changes in corneal curvature in eyes with progressive keratoconus or post-refractive surgery ectasia.

ELIGIBILITY:
Inclusion Criteria:

i. Age 14 years or older for keratoconus subjects since disease often begins at puberty, and 18 years or older for post-refractive surgery keratectasia and post-transplant patients

ii. Signed, dated, written informed consent

iii. Having documented ectasia on topography or tomography after previous refractive surgery OR progressive keratoconus defined as one or more of the following changes over a period of 24 months or less before randomization:

* An increase of at least 1.0 diopter in the steepest keratometry value (or sim K), or
* an increase of at least 1.0 diopter in regular astigmatism evaluated by subjective manifest refraction, or
* a myopic shift (decrease in the spherical equivalent) of at least 0.5 diopters on subjective refraction, or
* documented decrease in visual acuity associated with irregular astigmatism and topographic features of ectasia

iv. Have minimal preoperative corneal thickness of 375 microns or more, as measured in the office with epithelium not yet removed

v. For subjects with non-post refractive surgery keratoconus diagnosis only:

* 14 years or older to 55 years of age,
* axial topography consistent with keratoconus such as presence of abnormal central or paracentral steepening on the corneal topography map, or presence of one or more slit lamp findings associated with keratoconus, such as

  * Fleischer ring
  * Vogt striae
  * Corneal thinning
  * Corneal scarring

vi. For contact lens wearers only:

Removal of contact lenses for the required period of time prior to final screening refraction:

* Contact lens minimum discontinuation time two weeks for soft, extended wear, soft toric, and rigid gas permeable lenses

vii. For patients with post-refractive surgery keratectasia:

* History of excimer laser refractive surgery with increasing refractive astigmatism and corneal topographic or keratometric astigmatism of 0.5 or more, or a history of decreasing best spectacle corrected visual acuity associated with the presence of topography suggestive of keratoconus or pellucid marginal degeneration or abnormal higher order aberrations (especially coma) on the aberration mapping of the eye.

viii. For patients with corneal transplants:

* History of corneal transplant for keratoconus with documented increasing refractive astigmatism and corresponding topographic irregularity occurring at least one year after corneal transplantation, not attributable to transplant suture removal and occurring during the most recent two years.

Exclusion Criteria:

i. Patients with excessively thin corneas. (Intraoperative minimal corneal thickness in the swollen state with the epithelium removed must exceed 400 microns)

ii. Keratometric readings greater than 62D

iii. No evidence of keratoconus/keratectasia progression over the prior three years

iv. Age less than 55 years but under

* 14 years for keratoconus patients
* 18 years for post-refractive surgery keratectasia and post-transplant patients

  v. Previous ocular condition in the eye(s) to be treated that might, in the investigator's opinion, predispose to complications (such as history herpes simplex keratitis, corneal melt, perforated corneal ulcer, descemetocele, prior corneal damage from chemical injury, herpes zoster keratitis, nystagmus, corneal scarring that significantly impairs vision, pre-existing glaucoma, glaucoma suspect, Goldmann applanation pressure exceeding 23 mm Hg, cataract, history of uveitis, active ocular disease that might lead to infection, corneal endothelial cell count below 1800 cells per square millimeter)

vi. Patients with a systemic condition that, in the investigator's opinion, might predispose to complications (such as Down syndrome, autoimmune disease, pregnancy or nursing at the time of initial treatment, history of alcohol abuse, being immunocompromised, allergy to riboflavin or other study medications)

vii. Patients who are unwilling or unable to comply with the study regimen and doctor's advice

viii. Patients unwilling to discontinue wear of rigid contact lenses in the eye to be operated on for at least one month before baseline examination, and for the first six months post-operatively

ix. Patient unwilling to discontinue contact lenses prior to baseline exam: one week for soft lenses, two weeks for rigid or soft toric lenses

x. Pregnancy at the time of proposed crosslinking

xi. Known hypersensitivity to riboflavin

xii. Central corneal endothelial cell count below 1400 cells per square millimeter.

xiii. Presence of significant central corneal stromal scar

xiv. History of delayed wound healing

xv. Immunocompromised patient

xvi. History of connective tissue disease (such as systemic lupus erythematosus, rheumatoid arthritis)

xvii. History of glaucoma, a Goldmann applanation pressure measured in keratoconus evaluation of above 24, or glaucoma suspect, xviii. Significant existing cataract

xix. Macular degeneration or confluent drusen of Bruchs membrane

xx. Evidence of past or present herpes simplex of the cornea

Ages: 14 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 250 (Estimated)
Dates: Start 2011-03; Primary Completion 2014-03 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Change in corneal curvature | 6 months
  Measured by maximum keratometry (Kmax)

SECONDARY OUTCOMES:
corrected distance acuity | 6 months
  best spectacle corrected distance acuity
corneal endothelial cell count | 6 months
pachymetry | 6 months
  Minimal corneal thickness

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Epstein, MD, Principal Investigator — Mercy Center for Corrective Eye Surgery
Locations (1):
- Mercy Center for Corrective Eye Surgery, McHenry, Illinois, United States

REFERENCES:
- [Result] Caporossi A, Mazzotta C, Baiocchi S, Caporossi T. Long-term results of riboflavin ultraviolet a corneal collagen cross-linking for keratoconus in Italy: the Siena eye cross study. Am J Ophthalmol. 2010 Apr;149(4):585-93. doi: 10.1016/j.ajo.2009.10.021. Epub 2010 Feb 6. PMID 20138607
- [Result] Goldich Y, Marcovich AL, Barkana Y, Avni I, Zadok D. Safety of corneal collagen cross-linking with UV-A and riboflavin in progressive keratoconus. Cornea. 2010 Apr;29(4):409-11. doi: 10.1097/ICO.0b013e3181bd9f8c. PMID 20164744
- [Result] Wittig-Silva C, Whiting M, Lamoureux E, Lindsay RG, Sullivan LJ, Snibson GR. A randomized controlled trial of corneal collagen cross-linking in progressive keratoconus: preliminary results. J Refract Surg. 2008 Sep;24(7):S720-5. doi: 10.3928/1081597X-20080901-15. PMID 18811118
- [Result] Raiskup-Wolf F, Hoyer A, Spoerl E, Pillunat LE. Collagen crosslinking with riboflavin and ultraviolet-A light in keratoconus: long-term results. J Cataract Refract Surg. 2008 May;34(5):796-801. doi: 10.1016/j.jcrs.2007.12.039. PMID 18471635
- [Result] Mazzotta C, Traversi C, Baiocchi S, Sergio P, Caporossi T, Caporossi A. Conservative treatment of keratoconus by riboflavin-uva-induced cross-linking of corneal collagen: qualitative investigation. Eur J Ophthalmol. 2006 Jul-Aug;16(4):530-5. doi: 10.1177/112067210601600405. PMID 16952090
- [Result] Caporossi A, Baiocchi S, Mazzotta C, Traversi C, Caporossi T. Parasurgical therapy for keratoconus by riboflavin-ultraviolet type A rays induced cross-linking of corneal collagen: preliminary refractive results in an Italian study. J Cataract Refract Surg. 2006 May;32(5):837-45. doi: 10.1016/j.jcrs.2006.01.091. PMID 16765803
- See also: Educational material in website of Mercy Center for Corrective Eye Surgery — http://www.ICanSee.com